CLINICAL TRIAL: NCT02031185
Title: A Wearable mHealth Device to Promote Teenagers' Physical Activity: A Pilot RCT
Brief Title: A Wearable mHealth Device to Promote Teenagers' Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SCRI-24100018
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait-list control (No Intervention): No intervention
- FitBit only (Experimental): Participants will use the FitBit device
  Interventions: Behavioral: FitBit only
- FitBit and Text Messages (Experimental): Participants will use the FitBit device and receive daily affective text messages
  Interventions: Behavioral: FitBit and Text Messages

INTERVENTIONS:
Behavioral: FitBit only — Participants will use the FitBit device
  Arms: FitBit only
Behavioral: FitBit and Text Messages — Participants will use the FitBit device and receive daily affective text messages
  Arms: FitBit and Text Messages

SUMMARY:
Due to disparities in childhood obesity, interventions for physical activity promotion and obesity prevention for low socioeconomic and racial/ethnic minority children and adolescents are vital to address disparities across the lifespan. Mobile health applications (mHealth apps) are a rapidly growing and promising approach for interactive and individualized interventions for disease prevention. Smart phones are a promising platform to reach racial/ethnic minority and lower income groups due to high rates of adoption of smart phone usage among these groups When paired with wearable sensing devices, mHealth apps for smart phones can collect data and provide feedback to users in real time. In a study among university students regarding mHealth apps, participants expressed interest in the "ability to record and track behaviors and goals and the ability to acquire advice and information 'on the go'". For physical activity in particular, wearable physical activity monitors designed for consumers that objectively measure and display data related to an individual's physical activity on smart phones through mHealth apps have become widely available and affordable. These wearable devices wirelessly upload data and provide users with physical activity data visualization and goal setting features that can be customized for each user via internet-based applications for smart phones, tablets, and/or computers. While several internet-based behavioral programs to promote pediatric physical activity have been reported in a recent review, none examined wearable sensing devices coupled with mHealth apps. Similarly, a 2013 review on mHealth technologies for physical activity assessment and promotion reported no studies that used wearable sensing devices for intervention delivery and called for research to evaluate feasibility.

The Primary Goal is to conduct a pilot randomized controlled trial (RCT) of the FitBit Flex, a popular wearable physical activity sensing device that allows data visualization and goal setting on smart phones. The target population will be adolescents ages 14-18 years old in the Seattle-metro area (n=40) with approximately 50% from low income households or belonging to a racial/ethnic minority. We will target this older age group since they have the lowest levels of physical activity among the pediatric population. This pilot study will provide feasibility and preliminary data for a future R01-funded RCT of the Flex mHealth device and app.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old
* lives in the Seattle-metro area
* able to complete forms in English
* no restrictions by a health care provider on physical activity or walking
* own a smart phone or similar FitBit compatible mobile device (e.g. iPod Touch)
* agree to install and share data from the FitBit Flex smart phone app with the investigators
* attends study high school or health clinic or receives and clicks on a Facebook advertisement for the study

Exclusion Criteria:

* has been restricted by a health care provider for physical activity or walking
* does not live in the Seattle-metro area
* does not attend a study school or clinic, or did not receive a Facebook advertisement for the study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Post-intervention daily steps | Measured during weeks 3-4 of the intervention

SECONDARY OUTCOMES:
Pre-intervention daily steps | Baseline
Pre-intervention moderate-to-vigorous physical activity (MVPA) | Baseline
  Accelerometry
Post-intervention moderate-to-vigorous physical activity | During weeks 3-4 of the intervention
  accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, MD, MPH, Principal Investigator — University of Washington; Megan Moreno, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States